CLINICAL TRIAL: NCT06972771
Title: Trop2-targeting the Second Near-Infrared Fluorescence(NIR-II ) Molecular Probe for Guided Identification of Non-Muscle-Invasive Bladder Cancer
Brief Title: Trop2-targeting NIR-II Molecular Probe for Guided Identification of Non-Muscle-Invasive Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2024-304
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Non-Muscle-Invasive Bladder Cancer
Keywords: Trop2; NIR-II; Non-Muscle-Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TTP-ICG incubation: The resected clinical specimens will be completely soaked in the TTP-ICG incubation solution (5, 10, 20 μg/mL) for 3, 5, or 10 minutes, followed by 5 minutes of rinsing with PBST buffer and drying with absorbent paper. The NIR-II fluorescence imaging will be then performed under the DPM NIR-II system. And the correlation between pathological characterization and fluorescent information will be further analyzed.
  Interventions: Diagnostic Test: TTP-ICG incubation solution

INTERVENTIONS:
Diagnostic Test: TTP-ICG incubation solution — Clinical specimens will be incubated with TTP-ICG with different concentrations and times.

SUMMARY:
Bladder cancer ranks as the fourth most common malignancy among males the United States . Approximately 75% of patients present with non-muscle-invasive bladder cancer (NMIBC). For the diagnosis and treatment of NMIBC, current guidelines widely recommend white light cystoscopy (WLC) and transurethral resection of the bladder tumor (TURBT). Unfortunately, up to 70% of patients with NMIBC experience intravesical recurrence within five years of their initial treatment. The high recurrence rates necessitate long-term surveillance for most NMIBC patients, making it one of the most costly malignancies to manage. In fact, a higher risk of disease recurrence is also associated with the now widely used WLC and TURBT, which cause false-negative investigations with an inadequate resection or residual tumor, especially when urothelial tumors present as carcinoma in situ or multiple.

Indocyanine green (ICG)-based the second near-infrared (NIR-II) fluorescence imaging offers real-time visualization during surgery, potentially reducing residual tumor. Herein, the investigators will introduce a novel NIR-II probe, TTP-ICG, based on a Trop2-targeting peptide (TTP) and an approach which enables differentiation between cancer and para-cancer . In brief, tissues will be soaked in TTP-ICG after resection, and their histological characterization will be determined under NIR-II fluorescence imaging. Pathological confirmation will further validate our approach.

To explore the conditions for the future in vivo real-time identification of NMIBC during NIR-II fluorescence -guided surgery.

DETAILED DESCRIPTION:
After patient enrollment, surgical treatment will be administered based on clinical diagnosis and treatment. Following the surgery, excised tissues will undergo incubation with TTP-ICG following this specific procedure:

1. Preparation of the incubation solution: TTP-ICG will be dissolved in phosphate-buffered saline (PBS) at room temperature in the dark, with varying concentrations (5, 10, 20 μg/mL).
2. Incubation of the cancer and adjacent tissues: The excised tissues will be immersed and gently agitated in the incubation solution for 3, 5, or 10 minutes. Subsequently, they will be rinsed with PBST buffer (PBS with Tween 20) for 5 minutes and dried using absorbent paper.
3. Acquisition of NIR-II images: NIR-II images and fluorescent intensities will be captured using the " Digital Precision Medicine (DPM) " NIR-II system, optimized with appropriate parameters.
4. Pathological diagnosis and data analysis: Hematoxylin and eosin (H&E) staining, along with immuno-histochemistry (IHC) , will be performed. The subsequent correlation between pathological characterization and fluorescent information will be further analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-80 years of age
* Patients with suspected non-muscle-invasive bladder cancer scheduled to undergo surgical intervention.
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

* Patients unable to participate in the consent process
* Patients had contraindications to surgery, such as serious cardiopulmonary disease, coagulation dysfunction, etc
* Other conditions that the researcher considers inappropriate to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll 30 patients, who have been suspected non-muscle-invasive bladder cancer scheduled to undergo surgical intervention. Following the surgery, the resected tissues will be incubated with the TTP-ICG solution, and NIR-II fluorescence signals from the tissues will be collected.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Differentiation of bladder cancer and para-cancer tissues | 6 months
  NIR-II fluorescence intensity of bladder cancer and para-cancer tissues after TTP-ICG incubation : NIR-II fluorescence imaging acquisition and intensity analysis was conducted using the Digital Precision Medicine (DPM) NIR-II system. Following initial system parameter calibration and spatial scaling, fluorescence signals were captured and quantitatively analyzed to determine whether the tissue is benign or malignant through proprietary diagnostic algorithms.

SECONDARY OUTCOMES:
Correlation between NIR-Ⅱ fluorescence and pathological diagnosis of tissues | 6 months
  Examination of H&E pathological results and Trop2 IHC results in resected tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China